CLINICAL TRIAL: NCT07326761
Title: Microplastic Exposure in Neonates Receiving Parenteral Nutrition: A Prospective Cohort Study in the NICU
Acronym: Microplastics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huiyi Li (Other)
Responsible Party: Sponsor-Investigator, Huiyi Li, Deputy director of the nurse, the Second People's Hospital of Guangdong Province, Guangdong Second Provincial General Hospital
Organization: Guangdong Second Provincial General Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2025-KY-KZ-164-02
Record Dates: First submitted 2025-11-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Microplastics Exposure
Keywords: Microplastics; Parenteral Nutrition; newborns
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Long-term exposure group (Active Comparator): Premature infants requiring continuous parenteral nutrition support for over 14 days due to severe feeding difficulties, necrotizing enterocolitis (NEC), short bowel syndrome, or other serious intestinal diseases
  Interventions: Behavioral: No Intervention: Observational Cohort
- Short-term exposure group (Placebo Comparator): Premature infants receiving parenteral nutrition support for 3-7 days due to early adaptation issues (e.g., respiratory distress, temporary feeding intolerance) and having successfully transitioned to total parenteral nutrition for at least 48 hours prior to blood sample collection. This group represents common short-term iatrogenic exposure in NICU settings.
  Interventions: Behavioral: No Intervention: Observational Cohort
- Control group (No Intervention): The study included healthy full-term newborns born at 37 weeks or later gestational age. These infants received neither intravenous nutritional support nor planned fluid therapy, serving as baseline microplastic levels in the absence of iatrogenic exposure.

INTERVENTIONS:
Behavioral: No Intervention: Observational Cohort — These infants received neither intravenous nutritional support nor planned fluid therapy, serving as baseline microplastic levels in the absence of iatrogenic exposure.
  Arms: Long-term exposure group; Short-term exposure group

SUMMARY:
The purpose of this study is to explore a potential exposure risk in the neonatal intensive care unit, namely, the iatrogenic microplastic exposure that critically ill newborns may face when receiving life-saving parenteral nutrition (intravenous nutrition delivered through a plastic infusion system). Therefore, the investigators designed a prospective study. By comparing three groups of newborns-those requiring long-term intravenous nutrition, short-term intravenous nutrition, and no intravenous nutrition-and collecting blood samples with strictly contamination-proof non-plastic instruments, the investigators used high-precision Raman spectroscopy for detection. For the first time, they attempted to systematically and quantitatively analyze the microplastic load in neonatal blood and its relationship with the duration of intravenous nutrition. The aim of this study is to provide novel scientific evidence for evaluating microplastic exposure in the neonatal medical environment, with the ultimate goal of establishing a basis for developing safer clinical practices and medical material standards in the future, thereby better protecting the long-term health of vulnerable newborns.

DETAILED DESCRIPTION:
BACKGROUND: As a new environmental pollutant, microplastics has been found in many tissues of human body. Newborns, especially those who need intensive care and parenteral nutrition, may face a unique and persistent risk of microplastics exposure through plastic medical equipment, but their internal load is not clear.

Objective: The purpose of this study is to systematically evaluate the microplastics exposure of newborns in neonatal intensive care unit (NICU) during hospitalization through a prospective observation cohort, focusing on the potential relationship between the duration of parenteral nutrition and microplastics load.

Methods: Twelve newborns were recruited in 2025, and were divided into long-term exposure group, short-term exposure group and unexposed control group according to the support time of parenteral nutrition. In this study, blood samples of newborns were collected under strict pollution control, and microplastics in the samples was qualitatively and quantitatively analyzed by confocal micro-Raman spectroscopy.

ELIGIBILITY:
Inclusion criteria:

* Newborns hospitalized in neonatal intensive care unit of Guangdong Second People's Hospital in 2025.
* The gestational age of birth is ≥ 28 weeks.
* Intravenous nutrition time is 1-56 days.
* The mother has no serious basic diseases (such as heart disease, chronic kidney disease, mental illness, hypertension, diabetes, etc.).

Exclusion criteria:

* There are serious congenital malformations or chromosomal abnormalities. Combined with other serious diseases that may affect the metabolism or distribution of microplastics (such as congenital metabolic abnormality, liver or renal insufficiency).
* Parents or legal guardians withdraw informed consent.
* Death or automatic discharge within 72 hours after birth.

Ages: 1 Hour to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Particle number of neonatal blood sample | parenteral nutrition support for over 14 days，parenteral nutrition support for 3-7 days，The first day after birth
  The number of microplastics granules in newborn blood was detected.

SECONDARY OUTCOMES:
Education | Day 1
  questionnaire
Occupation | Day 1
  questionnaire
Annual income per capita (CNY) | Day 1
  questionnaire
Parity | Day 1
  questionnaire
Mode of conception | Day 1
  questionnaire
Birth outcome | Day 1
  questionnaire
Sex of newborns | Day 1
  physiological parameter
Mode of delivery | Day 1
  physiological parameter
Newborn weight (kg) | Day 1
  physiological parameter
Length of intravenous nutrition | Day 1
  physiological parameter

CONTACTS AND LOCATIONS:
Locations (1):
- The Second People's Hospital of Guangdong Province affiliated to Jinan University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT07326761/Prot_SAP_000.pdf
  • Informed Consent Form (2025-01-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT07326761/ICF_001.pdf